CLINICAL TRIAL: NCT06952192
Title: Effectiveness of Virtual Reality in Reducing Anxiety, Fear, and Pain in Pediatric Patients Undergoing Skin Prick Testing: A Cross-Over Study
Brief Title: Virtual Reality During Skin Prick Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Full Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 11n24
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Allergy
Keywords: virtual reality; skin prick test; pediatric allergy; anxiety; pain; compliance
MeSH Terms: conditions — Hypersensitivity; Anxiety Disorders; Pain; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental)
  Interventions: Device: Virtual reality
- Standard of care (No Intervention)

INTERVENTIONS:
Device: Virtual reality — VR application via a head-mounted display one minute before and throughout the SPT procedure. The VR intervention utilized a Samsung Gear VR headset (Samsung, Seoul, South Korea) in conjunction with a Samsung S7 or S8 mobile device to provide an immersive and engaging experience. Children were allowed to choose from a range of age-appropriate VR content designed to enhance engagement and relaxation. Prior to the procedure, children were trained on how to use the headset by study staff to ensure a smooth experience.
  Arms: Virtual reality

SUMMARY:
Skin prick testing (SPT) is a cornerstone diagnostic procedure for identifying allergic sensitizations in pediatric patients. Despite being minimally invasive, it often provokes considerable anxiety, fear, and pain, potentially compromising test accuracy due to poor compliance. Virtual Reality (VR) has emerged as a promising non-pharmacological tool for procedural distress management, yet its application in allergy diagnostics remains underexplored.

To evaluate the effectiveness of VR in reducing procedural anxiety, fear, and pain, and in improving compliance in children undergoing SPT.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed history of allergic symptoms related to either environmental or food allergens
* between 4 and 18 years of age

Exclusion Criteria:

* history of seizure disorders,
* motion sickness,
* severe developmental delay,
* non-Italian-speaking patients
* Participants who had used systemic antihistamines or corticosteroids within the past seven days

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
change of procedural anxiety in pediatric patients undergoing skin prick test | during the procedure
  The primary objective of this study was to evaluate the effectiveness of VR in reducing procedural anxiety in pediatric patients undergoing SPT. Anxiety levels were assessed using the CAM scale before (0), during (1), post procedure, i.e., one minute after the procedure (2).

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No